CLINICAL TRIAL: NCT03598205
Title: Combination Therapy Based on Curcumin and Intravitreal Dexamethasone in Diabetic Macular Edema Treatment to Help the Antiedemigenous Effect of Intravitreal Dexamethasone in Subjects With Diabetic Macular Edema (DME)
Brief Title: Curcumin and Intravitreal Dexamethasone in Diabetic Macular Edema
Acronym: DIABEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione G.B. Bietti, IRCCS (Other)
Responsible Party: Principal Investigator, Mariacristina Parravano, MD , Head RETINA UNIT, Fondazione G.B. Bietti, IRCCS
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FGBBietti
Record Dates: First submitted 2018-07-13; First posted 2018-07-26 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Macular Edema
Keywords: Therapy for diabetic macular edema; Curcumin formulation (DIABEC)

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DIABEC plus intravitreal dexamethazone (Experimental): Intervention:Curmin formulation (DIABEC) plus dexamethazone intravitreal injection. Oral curcumin formulation (DIABEC 2 tablets/die) in combination with Dexamethazone (0,7 mg) intravitral injection for diabetic macular edema treatment
  Interventions: Combination Product: DIABEC plus intravitreal dexamethazone
- dexamethazone intravitreal injection (No Intervention): Intervention: dexamethazone intravitreal injection (0,7 mg) in PRN for diabetic macular edema treatment monotherapy.

INTERVENTIONS:
Combination Product: DIABEC plus intravitreal dexamethazone — Patients with diabetic macular edema undergoing to intravitreal dexamethazone will be randomized to curcumin formulation (DIABEC)
  Other Names: Intravitreal dexamethazone
  Arms: DIABEC plus intravitreal dexamethazone

SUMMARY:
The aim of the study is to explore the effect of a curcumin formulation in combination to intravitreal dexamethasone therapy in patients with diabetic macular edema on morphological retinal characteristics and retreatment times.

DETAILED DESCRIPTION:
Patients with diagnosis of clinically significant diabetic macular edema, confirmed by fluorangiography and OCT, undergoing to intravitreal dexamethazone injection will be enrolled in the study.

Enrollment will take place according to the inclusion/exclusion criteria set by the protocol.

The enrolled patients will be randomized for the addition or not of the curcumin formulation (2 tablets/die for 6 months) to intravitreal therapy.

ELIGIBILITY:
Inclusion Criteria:

* - Patients with clinically significant diabetic macular edema in non-proliferative diabetic retinopathy, diagnosed by fluorangiography and OCT
* Naive patients
* Patients with clinically significant DME who have not been treated for more than 3 months with anti-VEGF therapy and for more than 6 months with intravitreal injection of dexamethasone
* Central retinal thickness (CRT) at OCT> 300 microns
* Best Corrected Visual Acuity (BCVA) with ETDRS tables at 4 meters not <20/400
* Ability to provide written informed consent and follow the procedures of the study

Exclusion Criteria:

* Retinal pathologies other than diabetic macular edema
* Proliferative diabetic retinopathy
* Opacities that limit the execution and interpretation of diagnostic tests
* Surgical interventions in the study eye in the 3 months prior to the start of treatment
* Pregnancy
* Feeding time

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Mean difference in CRT from baseline to 6 months | 6 months
  To explore the effect of curcumin formulation in addition to intravitreal dexamethasone therapy on OCT central retinal thickness after 6 months of therapy

SECONDARY OUTCOMES:
Mean difference in BCVA from baseline to 6 months | 6 months
  To explore the effect of curcumin formulation in addition to intravitreal dexamethasone therapy on BCVA after 6 months of therapy
Evaluation of safety: incidence of Treatment-Emergent Adverse Events | 6 months
  To explore the safety of curcumin formulation (incidence of Treatment-Emergent Adverse Events ) in addition to intravitreal dexamethasone therapy after 6 months
Retreatment times | 6 months
  To explore the effect of curcumin formulation in addition to intravitreal dexamethasone therapy on retreatment times

CONTACTS AND LOCATIONS:
Overall Officials: Mariacristina Parravano, Principal Investigator — Fondazione G.B. Bietti, IRCCS
Locations (3):
- Italy (3):
  - Università Humanitas Gavazzeni Bergamo, Bergamo
  - Università degli Studi Magna Graecia, Catanzaro
  - Fondazione G.B.Bietti-IRCCS, Rome

IPD SHARING:
Plan to Share IPD: Undecided